CLINICAL TRIAL: NCT06036680
Title: Long-term Follow-up ProtDilat Study; Comparative Prospective Multicenter Randomized Study of Endoscopic Treatment of Stenosis in Crohn´s Disease: Self-expandable Metal Stent vs. Endoscopic Balloon Dilatation
Brief Title: Long-term Study of Endoscopic Treatment of Stenosis in Crohn´s Disease
Acronym: Long-ProtDilat
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: Clínica Girona (Unknown); Complejo Hospitalario Universitario de Vigo (Other); Consorcio Hospital Universitario Clinico de Valencia (Unknown); Hospital Clinic of Barcelona (Other); Hospital Comarcal de Inca (Other); Hospital de Terrassa (Other); Hospital General la Mancha-Centro (Unknown); Parc Taulí Hospital Universitari (Other); Hospital Universitario Ramón y Cajal (Unknown); Hospital Universitario Reina Sofía (Unknown); Hospital Universitari de Bellvitge (Other); University Hospital of Girona Dr. Josep Trueta (Network); Hospital Universitario La Fe (Other); Hospital Universitari Arnau de Vilanova (Unknown); Hospital Universitario de Burgos (Other); Hospital Universitario de Cáceres (Unknown); Hospital Universitario La Paz (Other); Hospital Universitario Rio Hortega (Unknown)
Responsible Party: Sponsor
Other Study IDs: Long-ProtDilat 1
Record Dates: First submitted 2023-09-04; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Crohn Disease; Stenosis
Keywords: endoscopic balloon dilatation; self-expanding metal stent
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic balloon dilatation (EBD) treated CD patients
- Self-expandable metal stent (SEMS) treated CD patients

SUMMARY:
Stenosis is one of the most frequent complications in patients with Crohn's disease (CD), causing greater morbidity and increasing the probability of repeated surgery and short bowel syndrome. Several endoscopic techniques, as an alternative to surgery, have been used in the treatment of fibrostenotic CD, with similar efficacy and lower risk of complications.

The ProtDilat study (NCT02395354) showed that both endoscopic balloon dilation (EBD) and self-expandable metal stents (SEMS) are efficient and safe for the treatment of stenosis in CD, while EBD shows therapeutic superiority (80.5 vs 51.3 %) at one year follow-up. However, this difference was not observed in the subanalysis of patients with stenosis > 3 cm (EBD: 66.7% vs SEMS: 63.6%) but with a lower cost for EBD (EDB 1,365.63 euros versus SEMS 1,923.55 euros).

Therefore, SEMS could be a suitable treatment option for longer stenoses in which EBD has proven to be less efficacious. Moreover, the long-term efficacy of both endoscopic treatments is still debated with scare information and without data from a clinical trial.

The aim of this study is to assess the long-term efficacy of EBD and SEMS, through the follow-up of the patients included in the ProtDilat study, being the primary objective of the study the percentage of patients free of surgical intervention at the end of follow-up. Retrospective study based on data from the ProtDilat trial (patients with CD, obstructive symptoms, with stenosis < 10cm). Data on medical, endoscopic and surgical treatment and smoking habits are collected.

ELIGIBILITY:
Inclusion Criteria:

* Age18-75.
* CD with predominating de novo and/or anastomotic fibrotic stenosis confirmed by endoscopy and radiology and accessible by endoscopy (colonoscopy).
* Stenosis previously treated with a stent and/or dilatation and with at least one year asymptomatic.
* Intestinal occlusion or sub-occlusion symptomatology.
* Refractoriness to conventional medical treatment (no response to accelerated step-up of normal therapeutic scale).
* Stenosis length < 10 cm.
* Maximum 2 stenoses.
* Informed consent of patient.

Exclusion Criteria:

* No informed consent of patient.
* Stenosis complicated by abscess, fistula, or important activity associated with CD not limited to the stenosis area.
* Stenosis previously treated with a stent and/or dilatation and with less than one year asymptomatic.
* Pregnancy or lactation.
* Any clinical condition that prevents the performance of endoscopy.
* Stenosis inaccessible by colonoscopy.
* No obstructive symptoms.
* Stenosis length ≥ 10 cm.
* Presenting more than 2 stenoses.
* Serious coagulation disorder (platelets < 70000; INR > 1.5)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CD patients included in the ProtDilat study that finished the follow-up
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of surgery-free patients post-treatment | end of long-term follow up (median 7 years post-treatment)

SECONDARY OUTCOMES:
Percentage of patients that have not required any endoscopic retreatment | end of long-term follow up (median 7 years post-treatment)
Long-term effectiveness of endoscopic treatment (SEMS vs EBD): percentage of patients free of surgery and who have not required any endoscopic retreatment | end of long-term follow up (median 7 years post-treatment)
Percentage of patients with safety issues and/or complications related to endoscopic or surgical treatment | end of long-term follow up (median 7 years post-treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Cosnes J, Gower-Rousseau C, Seksik P, Cortot A. Epidemiology and natural history of inflammatory bowel diseases. Gastroenterology. 2011 May;140(6):1785-94. doi: 10.1053/j.gastro.2011.01.055. PMID 21530745
- [Background] Peyrin-Biroulet L, Loftus EV Jr, Colombel JF, Sandborn WJ. The natural history of adult Crohn's disease in population-based cohorts. Am J Gastroenterol. 2010 Feb;105(2):289-97. doi: 10.1038/ajg.2009.579. Epub 2009 Oct 27. PMID 19861953
- [Background] Solberg IC, Vatn MH, Hoie O, Stray N, Sauar J, Jahnsen J, Moum B, Lygren I; IBSEN Study Group. Clinical course in Crohn's disease: results of a Norwegian population-based ten-year follow-up study. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1430-8. doi: 10.1016/j.cgh.2007.09.002. PMID 18054751
- [Background] Shen B, Kochhar G, Navaneethan U, Liu X, Farraye FA, Gonzalez-Lama Y, Bruining D, Pardi DS, Lukas M, Bortlik M, Wu K, Sood A, Schwartz DA, Sandborn WJ; Global Interventional Inflammatory Bowel Disease Group. Role of interventional inflammatory bowel disease in the era of biologic therapy: a position statement from the Global Interventional IBD Group. Gastrointest Endosc. 2019 Feb;89(2):215-237. doi: 10.1016/j.gie.2018.09.045. Epub 2018 Oct 24. PMID 30365985
- [Background] Loras C, Manosa M, Andujar X, Sanchiz V, Marti-Gallostra M, Zabana Y, Gutierrez A, Barreiro-de Acosta M; en representacion de GETECCU. Position Statement. Recommendations of the Spanish Group on Crohn's Disease and Ulcerative Colitis (GETECCU) on the treatment of strictures in Crohn's disease. Gastroenterol Hepatol. 2022 Apr;45(4):315-334. doi: 10.1016/j.gastrohep.2021.07.001. Epub 2021 Jul 15. English, Spanish. PMID 34274357
- [Background] Bettenworth D, Gustavsson A, Atreja A, Lopez R, Tysk C, van Assche G, Rieder F. A Pooled Analysis of Efficacy, Safety, and Long-term Outcome of Endoscopic Balloon Dilation Therapy for Patients with Stricturing Crohn's Disease. Inflamm Bowel Dis. 2017 Jan;23(1):133-142. doi: 10.1097/MIB.0000000000000988. PMID 28002130
- [Background] Hassan C, Zullo A, De Francesco V, Ierardi E, Giustini M, Pitidis A, Taggi F, Winn S, Morini S. Systematic review: Endoscopic dilatation in Crohn's disease. Aliment Pharmacol Ther. 2007 Dec;26(11-12):1457-64. doi: 10.1111/j.1365-2036.2007.03532.x. Epub 2007 Sep 28. PMID 17903236
- [Background] Morar PS, Faiz O, Warusavitarne J, Brown S, Cohen R, Hind D, Abercrombie J, Ragunath K, Sanders DS, Arnott I, Wilson G, Bloom S, Arebi N; Crohn's Stricture Study (CroSS) Group. Systematic review with meta-analysis: endoscopic balloon dilatation for Crohn's disease strictures. Aliment Pharmacol Ther. 2015 Nov;42(10):1137-48. doi: 10.1111/apt.13388. Epub 2015 Sep 11. PMID 26358739
- [Background] Navaneethan U, Lourdusamy V, Njei B, Shen B. Endoscopic balloon dilation in the management of strictures in Crohn's disease: a systematic review and meta-analysis of non-randomized trials. Surg Endosc. 2016 Dec;30(12):5434-5443. doi: 10.1007/s00464-016-4902-1. Epub 2016 Apr 28. PMID 27126619
- [Background] Thienpont C, D'Hoore A, Vermeire S, Demedts I, Bisschops R, Coremans G, Rutgeerts P, Van Assche G. Long-term outcome of endoscopic dilatation in patients with Crohn's disease is not affected by disease activity or medical therapy. Gut. 2010 Mar;59(3):320-4. doi: 10.1136/gut.2009.180182. Epub 2009 Oct 19. PMID 19840991
- [Background] Gustavsson A, Magnuson A, Blomberg B, Andersson M, Halfvarson J, Tysk C. Endoscopic dilation is an efficacious and safe treatment of intestinal strictures in Crohn's disease. Aliment Pharmacol Ther. 2012 Jul;36(2):151-8. doi: 10.1111/j.1365-2036.2012.05146.x. Epub 2012 May 22. PMID 22612326
- [Background] Atreja A, Aggarwal A, Dwivedi S, Rieder F, Lopez R, Lashner BA, Brzezinski A, Vargo JJ, Shen B. Safety and efficacy of endoscopic dilation for primary and anastomotic Crohn's disease strictures. J Crohns Colitis. 2014 May;8(5):392-400. doi: 10.1016/j.crohns.2013.10.001. Epub 2013 Nov 1. PMID 24189349
- [Background] Andujar X, Loras C, Gonzalez B, Socarras M, Sanchiz V, Bosca M, Domenech E, Calafat M, Rodriguez E, Sicilia B, Calvet X, Barrio J, Guardiola J, Iglesias E, Casanova MJ, Ber Y, Monfort D, Lopez-Sanroman A, Rodriguez-Lago I, Bujanda L, Marquez L, Martin-Arranz MD, Zabana Y, Fernandez-Banares F, Esteve M; ENEIDA registry of GETECCU. Efficacy and safety of endoscopic balloon dilation in inflammatory bowel disease: results of the large multicenter study of the ENEIDA registry. Surg Endosc. 2020 Mar;34(3):1112-1122. doi: 10.1007/s00464-019-06858-z. Epub 2019 May 29. PMID 31144122
- [Background] Attar A, Maunoury V, Vahedi K, Vernier-Massouille G, Vida S, Bulois P, Colombel JF, Bouhnik Y; GETAID. Safety and efficacy of extractible self-expandable metal stents in the treatment of Crohn's disease intestinal strictures: a prospective pilot study. Inflamm Bowel Dis. 2012 Oct;18(10):1849-54. doi: 10.1002/ibd.22844. Epub 2011 Dec 11. PMID 22161935
- [Background] Levine RA, Wasvary H, Kadro O. Endoprosthetic management of refractory ileocolonic anastomotic strictures after resection for Crohn's disease: report of nine-year follow-up and review of the literature. Inflamm Bowel Dis. 2012 Mar;18(3):506-12. doi: 10.1002/ibd.21739. Epub 2011 May 3. PMID 21542067
- [Background] Loras C, Perez-Roldan F, Gornals JB, Barrio J, Igea F, Gonzalez-Huix F, Gonzalez-Carro P, Perez-Miranda M, Espinos JC, Fernandez-Banares F, Esteve M. Endoscopic treatment with self-expanding metal stents for Crohn's disease strictures. Aliment Pharmacol Ther. 2012 Nov;36(9):833-9. doi: 10.1111/apt.12039. PMID 22966851
- [Background] Loras C. Endoscopic Stenting for Inflammatory Bowel Disease Strictures. Gastrointest Endosc Clin N Am. 2022 Oct;32(4):699-717. doi: 10.1016/j.giec.2022.04.004. PMID 36202511
- [Background] Loras C, Andujar X, Gornals JB, Sanchiz V, Brullet E, Sicilia B, Martin-Arranz MD, Naranjo A, Barrio J, Duenas C, Foruny JR, Busquets D, Monfort D, Pineda JR, Gonzalez-Huix F, Perez-Roldan F, Pons V, Gonzalez B, Reyes Moreno J, Sainz E, Guardiola J, Bosca-Watts MM, Fernandez-Banares F, Mayor V, Esteve M; Grupo Espanol de Trabajo de la Enfermedad de Crohn y Colitis Ulcerosa (GETECCU). Self-expandable metal stents versus endoscopic balloon dilation for the treatment of strictures in Crohn's disease (ProtDilat study): an open-label, multicentre, randomised trial. Lancet Gastroenterol Hepatol. 2022 Apr;7(4):332-341. doi: 10.1016/S2468-1253(21)00386-1. Epub 2022 Jan 20. PMID 35065738
- [Background] Ding NS, Yip WM, Choi CH, Saunders B, Thomas-Gibson S, Arebi N, Humphries A, Hart A. Endoscopic Dilatation of Crohn's Anastomotic Strictures is Effective in the Long Term, and Escalation of Medical Therapy Improves Outcomes in the Biologic Era. J Crohns Colitis. 2016 Oct;10(10):1172-8. doi: 10.1093/ecco-jcc/jjw072. Epub 2016 Mar 12. PMID 26971054
- [Background] Takeda T, Kishi M, Takatsu N, Takada Y, Beppu T, Miyaoka M, Hisabe T, Ueki T, Arima H, Hirai F, Yao K. Long-term outcomes of endoscopic balloon dilation for intestinal strictures in patients with Crohn's disease during maintenance treatment with anti-tumor necrosis factor alpha antibodies. Dig Endosc. 2022 Mar;34(3):517-525. doi: 10.1111/den.14073. Epub 2021 Jul 18. PMID 34185921
- [Background] Sivasailam B, Lane BF, Cross RK. Endoscopic Balloon Dilation of Strictures: Techniques, Short- and Long-Term Outcomes, and Complications. Gastrointest Endosc Clin N Am. 2022 Oct;32(4):675-686. doi: 10.1016/j.giec.2022.04.006. Epub 2022 Sep 7. PMID 36202509
- [Background] Lian L, Stocchi L, Remzi FH, Shen B. Comparison of Endoscopic Dilation vs Surgery for Anastomotic Stricture in Patients With Crohn's Disease Following Ileocolonic Resection. Clin Gastroenterol Hepatol. 2017 Aug;15(8):1226-1231. doi: 10.1016/j.cgh.2016.10.030. Epub 2016 Nov 2. PMID 27816758
- [Background] Wang X, Xia H, Liu S, Cao L, You F. Epigenetic regulation in antiviral innate immunity. Eur J Immunol. 2021 Jul;51(7):1641-1651. doi: 10.1002/eji.202048975. Epub 2021 May 27. PMID 33964027